CLINICAL TRIAL: NCT00011648
Title: Determining the Prevalence and Prognosis of Secondary Pulmonary Hypertension in Adult Patients With Sickle Cell Anemia
Brief Title: Secondary Pulmonary Hypertension in Adults With Sickle Cell Anemia
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010088; 01-H-0088
Record Dates: First submitted 2001-02-24; First posted 2001-02-26 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12-15

CONDITIONS: Pulmonary Hypertension; Sickle Cell Anemia; Sickle Cell Disease
Keywords: Echocardiogram; Morbidity; Mortality; Natural History; Sickle Cell Anemia; Secondary Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-SCD: 200 Men and Women without a diagnosis of sickle cell disease 18 years of age or older
- SCD: 1000 Men and Women with a diagnosis of sickle cell disease

SUMMARY:
The purpose of this study is to determine how often people with sickle cell anemia develop pulmonary hypertension a serious disease in which blood pressure in the artery to the lungs is elevated.

Men and women 18 years of age and older with sickle cell anemia may be eligible for this study. Participants will undergo an evaluation at Howard University s Comprehensive Sickle Cell Center in Washington, D.C. or at the National Institutes of Health in Bethesda, Maryland. It will include the following:

* medical history
* physical examination
* blood collection (no more than 50 ml., or about 1/3 cup) to confirm the diagnosis of sickle cell anemia, sickle cell trait or beta-thalassemia (Some blood will be stored for future research testing on sickle cell anemia.)
* echocardiogram (ultrasound test of the heart) to check the pumping action of the heart and the rate at which blood travels through the tricuspid valve.

Following this evaluation, a study nurse will contact participants twice a month for 2 months and then once every 3 months for the next 3 years for a telephone interview. The interview will include questions about general health and recent health-related events, such as hospitalizations or emergency room visits.

DETAILED DESCRIPTION:
Sickle cell anemia is an autosomal recessive disorder and the most common genetic disease affecting African-Americans. Approximately 0.15% of African-Americans are homozygous for sickle cell disease, and 8% have sickle cell trait. Acute pain crisis, acute chest syndrome (ACS), and secondary pulmonary hypertension are common complications of sickle cell anemia. Mortality rates of sickle cell patients with pulmonary hypertension are significantly increased as compared to patients without pulmonary hypertension. Recent studies report up to 40% mortality at 22 months after detection of elevated pulmonary artery pressures in sickle cell patients. Furthermore, pulmonary hypertension is thought to occur in up to 30% of clinic patients with sickle cell anemia.

This study is designed to determine the prevalence and prognosis of secondary pulmonary hypertension in adult patients with sickle cell anemia, and to determine whether genetic polymorphisms in candidate genes contribute to its development or response to treatment.

ELIGIBILITY:
* INCLUSION CRITERIA FOR SICKLE CELL PATIENTS:
* Male and females over 18 years of age.
* Diagnosis of sickle cell disease (electrophoretic documentation of SS, SC, or S-beta thallassemia genotype is required).

EXCLUSION CRITERIA FOR SICKLE CELL PATIENTS:

* Hb A-only phenotype and sickle cell trait.
* Decisionally impaired subjects.
* Pregnant or lactating women

INCLUSION CRITERIA FOR CONTROL SUBJECTS:

* Male and females African American subjects over 18 years of age.
* Exclusion of sickle cell disease (electrophoretic documentation of hemoglobin A is required).

EXCLUSION CRITERIA FOR CONTROL SUBJECTS:

* Diagnosis of sickle cell disease (electrophoretic documentation of SS, or SC, or SB thallassemia genotype is required.)
* Decisionally impaired subjects.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and females African American subjects over 18 years of age. Exclusion of sickle cell disease (electrophoretic documentation of hemoglobin A is required)
Sampling Method: Non-Probability Sample
Enrollment: 986 (Actual)
Dates: Start 2008-02-19 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence and prognosis of secondary pulmonary hypertension in adult patients with sickle cell anemia. | 10 years
  predictive of any clinical outcome or response in sickle cell disease will provide preliminary evidence for further investigation

SECONDARY OUTCOMES:
To determine whether genetic polymorphisms in candidate genes contribute to its development or response to treatment. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Howard University Hospital, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Derived] Parrow NL, Doherty JM, Conrey A, Thein SL, Fleming RE. Relationships Between Markers of Iron Status and Hematological Parameters in Patients With Sickle Cell Disease. Adv Hematol. 2024 Dec 3;2024:9872440. doi: 10.1155/ah/9872440. eCollection 2024. PMID 39659429
- [Derived] van Vuren AJ, Minniti CP, Mendelsohn L, Baird JH, Kato GJ, van Beers EJ. Lactate dehydrogenase to carboxyhemoglobin ratio as a biomarker of heme release to heme processing is associated with higher tricuspid regurgitant jet velocity and early death in sickle cell disease. Am J Hematol. 2021 Sep 1;96(9):E315-E318. doi: 10.1002/ajh.26243. Epub 2021 Jun 10. No abstract available. PMID 34000072
- [Derived] Sachdev V, Tian X, Gu Y, Nichols J, Sidenko S, Li W, Beri A, Layne WA, Allen D, Wu CO, Thein SL. A phenotypic risk score for predicting mortality in sickle cell disease. Br J Haematol. 2021 Mar;192(5):932-941. doi: 10.1111/bjh.17342. Epub 2021 Jan 28. PMID 33506990
- [Derived] Nguyen KL, Tian X, Alam S, Mehari A, Leung SW, Seamon C, Allen D, Minniti CP, Sachdev V, Arai AE, Kato GJ. Elevated transpulmonary gradient and cardiac magnetic resonance-derived right ventricular remodeling predict poor outcomes in sickle cell disease. Haematologica. 2016 Feb;101(2):e40-3. doi: 10.3324/haematol.2015.125229. Epub 2015 Nov 20. No abstract available. PMID 26589907
- [Derived] Fitzhugh CD, Hsieh MM, Allen D, Coles WA, Seamon C, Ring M, Zhao X, Minniti CP, Rodgers GP, Schechter AN, Tisdale JF, Taylor JG 6th. Hydroxyurea-Increased Fetal Hemoglobin Is Associated with Less Organ Damage and Longer Survival in Adults with Sickle Cell Anemia. PLoS One. 2015 Nov 17;10(11):e0141706. doi: 10.1371/journal.pone.0141706. eCollection 2015. PMID 26576059
- [Derived] Wallen GR, Minniti CP, Krumlauf M, Eckes E, Allen D, Oguhebe A, Seamon C, Darbari DS, Hildesheim M, Yang L, Schulden JD, Kato GJ, Taylor JG 6th. Sleep disturbance, depression and pain in adults with sickle cell disease. BMC Psychiatry. 2014 Jul 21;14:207. doi: 10.1186/1471-244X-14-207. PMID 25047658
- [Derived] Darbari DS, Wang Z, Kwak M, Hildesheim M, Nichols J, Allen D, Seamon C, Peters-Lawrence M, Conrey A, Hall MK, Kato GJ, Taylor JG 6th. Severe painful vaso-occlusive crises and mortality in a contemporary adult sickle cell anemia cohort study. PLoS One. 2013 Nov 5;8(11):e79923. doi: 10.1371/journal.pone.0079923. eCollection 2013. PMID 24224021
- [Derived] Nekhai S, Xu M, Foster A, Kasvosve I, Diaz S, Machado RF, Castro OL, Kato GJ, Taylor JG 6th, Gordeuk VR. Reduced sensitivity of the ferroportin Q248H mutant to physiological concentrations of hepcidin. Haematologica. 2013 Mar;98(3):455-63. doi: 10.3324/haematol.2012.066530. Epub 2012 Oct 12. PMID 23065513
- [Derived] Minniti CP, Taylor JG 6th, Hildesheim M, O'Neal P, Wilson J, Castro O, Gordeuk VR, Kato GJ. Laboratory and echocardiography markers in sickle cell patients with leg ulcers. Am J Hematol. 2011 Aug;86(8):705-8. doi: 10.1002/ajh.22065. Epub 2011 May 31. PMID 21630312
- [Derived] Sundaram N, Tailor A, Mendelsohn L, Wansapura J, Wang X, Higashimoto T, Pauciulo MW, Gottliebson W, Kalra VK, Nichols WC, Kato GJ, Malik P. High levels of placenta growth factor in sickle cell disease promote pulmonary hypertension. Blood. 2010 Jul 8;116(1):109-12. doi: 10.1182/blood-2009-09-244830. Epub 2010 Mar 24. PMID 20335221
- [Derived] Kato GJ, Wang Z, Machado RF, Blackwelder WC, Taylor JG 6th, Hazen SL. Endogenous nitric oxide synthase inhibitors in sickle cell disease: abnormal levels and correlations with pulmonary hypertension, desaturation, haemolysis, organ dysfunction and death. Br J Haematol. 2009 May;145(4):506-13. doi: 10.1111/j.1365-2141.2009.07658.x. Epub 2008 Mar 17. PMID 19344390
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-H-0088.html